CLINICAL TRIAL: NCT01114516
Title: Role in Emergent Cerclage of Indomethacin and Antibiotics
Brief Title: Multifactorial Approach to Emergent Cerclage
Acronym: RECIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, William Grobman, principal investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00019610
Record Dates: First submitted 2010-04-29; First posted 2010-05-03 (Estimated); Results first posted 2014-10-10 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Cervical Insufficiency
Keywords: cervical insufficiency
MeSH Terms: conditions — Uterine Cervical Incompetence | interventions — Indomethacin; Anti-Bacterial Agents; Cefazolin; Clindamycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (No Intervention): emergent cerclage with no peri-operative antibiotics or indomethacin
- indomethacin and antibiotics (Experimental): perioperative antibiotics and indomethacin
  Interventions: Drug: Indomethacin and antibiotics (cefazolin or clindamycin)

INTERVENTIONS:
Drug: Indomethacin and antibiotics (cefazolin or clindamycin) — q8hr dosing of po indomethacin 50mg X 24 hrs and q8 hr 1 g IV cefazolin or 600 mg IV clindamycin
  Other Names: indocin, cleocin, ancef
  Arms: indomethacin and antibiotics

SUMMARY:
Though cervical insufficiency is a common cause of second trimester pregnancy loss, the placement of an emergent cerclage in these patients is thought to improve perinatal outcomes. It is unknown whether the use of tocolytics and antibiotics prolongs pregnancies complicated by need for emergent cerclage.

The objective is to determine whether administration of peri-operative antibiotics and indomethacin to patients receiving emergent cerclages for cervical insufficiency increases latency period to delivery compared with patients receiving emergent cerclage alone.

ELIGIBILITY:
Inclusion Criteria:

* GA 16+0 to 23+6 weeks
* Singleton gestation
* Presence of cervical dilation as diagnosed on digital examination
* Intact membranes

Exclusion Criteria:

* Age <18 years
* Allergy to NSAIDs
* Renal disease
* Allergy to penicillins AND clindamycin
* Currently on antibiotics or indomethacin for any reason
* HIV positive
* Pregnancies complicated by fetal congenital anomalies
* Preterm premature rupture of membranes
* Fever of 100.4 degrees Fahrenheit or higher
* Any patient having received a therapeutic cerclage during the current pregnancy

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2010-03; Primary Completion 2013-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Prentice Women's Hospital, Chicago, Illinois, United States

REFERENCES:
- [Result] Miller ES, Grobman WA, Fonseca L, Robinson BK. Indomethacin and antibiotics in examination-indicated cerclage: a randomized controlled trial. Obstet Gynecol. 2014 Jun;123(6):1311-1316. doi: 10.1097/AOG.0000000000000228. PMID 24807330

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Indomethacin and Antibiotics
Started | 26 | 27
Completed | 24 | 26
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Indomethacin and Antibiotics | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.7 (4.9) | 31.9 (6.5) | 30.3 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 26 | 50
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Gestational Latency Achieved Between Cerclage Placement and Time of Delivery
Description: Median gestational latency achieved Between Cerclage Placement and Time of Delivery
Time Frame: 24 weeks
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Control | Indomethacin and Antibiotics
Number analyzed (Participants) | 24 | 26
days | 80 [15 to 122] | 97 [57 to 125]
Statistical Analysis 1: Comparison: Control vs Indomethacin and Antibiotics; Kaplan Meier survival analysis; Test type: Superiority or Other; p = 0.018, Log Rank

2. Secondary Outcome: Gestational Latency of More Than 28 Days
Description: The frequency of achieving a gestational latency of more than 28 days
Time Frame: 28 days postpartum
Measure: Number; unit: percentage of participants
Arm/Group | Control | Indomethacin and Antibiotics
Number analyzed (Participants) | 24 | 26
percentage of participants | 62.5 | 92.3
Statistical Analysis 1: Comparison: Control vs Indomethacin and Antibiotics; Test type: Superiority or Other; Risk Ratio (RR) = 1.48, 95% CI 2-sided [1.06 to 2.05]

3. Secondary Outcome: Gestational Age at Delivery
Description: Median gestational age at delivery
Time Frame: 24 weeks
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Control | Indomethacin and Antibiotics
Number analyzed (Participants) | 24 | 26
weeks | 31.1 [22.9 to 38.5] | 34.8 [27.1 to 38.4]
Statistical Analysis 1: Comparison: Control vs Indomethacin and Antibiotics; Test type: Superiority or Other; p = 0.393, Kruskal-Wallis

4. Secondary Outcome: Neonatal Morbidity and Mortality
Description: Days spent in the neonatal intensive care unit
Time Frame: 1 year
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Control | Indomethacin and Antibiotics
Number analyzed (Participants) | 24 | 26
days | 95 [11 to 112] | 43 [19 to 107]

5. Secondary Outcome: Birthweight
Description: Median birthweight
Time Frame: 24 weeks
Measure: Median (Inter-Quartile Range); unit: grams
Arm/Group | Control | Indomethacin and Antibiotics
Number analyzed (Participants) | 24 | 26
grams | 2488 [955 to 3175] | 2850 [1440 to 3380]

ADVERSE EVENTS:
Arm/Group | Control | Indomethacin and Antibiotics
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/26
Other Adverse Events (participants affected / at risk) | 0/24 | 0/26

LIMITATIONS AND CAVEATS:
Because this study was not adequately powered to detect differences in perinatal outcomes, whether this adjunctive therapy affects these outcomes remains uncertain.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No